CLINICAL TRIAL: NCT01215448
Title: Impact of Wheatgrass Juice and Lifestyle Recommendations on Cancer Patients' Quality of Life During Chemotherapy Treatment
Brief Title: Wheatgrass Juice / Lifestyle Recommendations / Cancer Patients' Quality of Life / Chemotherapy Treatment
Acronym: 4001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, integrative Oncology Program, Medical director, The Oncology Service and Lin Medical center, Clalit Health Services., Carmel Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMC-10-0054-CTIL
Record Dates: First submitted 2010-09-28; First posted 2010-10-06 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Fatigue
Keywords: Fatigue; Quality of life; Lifestyle; Complementary medicine
MeSH Terms: conditions — Fatigue | interventions — Flour

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle changes (No Intervention): Lifestyle changes(booklet and audio cassette of recommended diet, physical activity and breathing exercises)
- Wheatgrass juice & lifestyle changes (Experimental): Wheatgrass juice & lifestyle changes
  Interventions: Dietary Supplement: Wheatgrass juice

INTERVENTIONS:
Dietary Supplement: Wheatgrass juice — 110 CC daily od frozen wheatgrass juice in the intervention arm
  Other Names: Triticum aestivum
  Arms: Wheatgrass juice & lifestyle changes

SUMMARY:
This study is aimed to study the impact of wheatgrass juice and lifestyle recommendations (diet, physical activity and breathing exercises) on the well being, fatigue and hematological parameters of chemotherapy-naive patients with no evidence for symptoms of active oncological disease.The researchers hypothesize that both wheatgrass juice and lifestyle recommendations can improve patient's well-being during chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy-naive patients will be offered to participate in a two arms study. Following consent, patients will be randomized to one of two arms. Patients in both arms will be provided by booklet and audio-cassette that specify lifestyle recommendations (diet, physical activity and breathing exercises). Patients in one of the study arms will be provided in addition with frozen wheatgrass juice (recommended daily dosage of 55-110 CC daily). Patients in both arms will be asked to fill in a daily patient's diary monitoring the practice of the lifestyle recommendations.

Baseline assessment will include the following questionnaires: ESAS, MYCAW, FACIT- Fatigue. Evaluation will include weekly ESAS and FACIT-Fatigue questionnaire and subsequent evaluation (including ESAS, MYCAW, FACIT- Fatigue questionnaires) following 3 and 4 chemotherapy cycles of treatment. Follow-up evaluation will be performed at the completion of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cancer with no sign of active disease
* First-time treatment with chemotherapy

Exclusion Criteria:

* Treatment with per os administration of chemotherapy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Assessing impact of wheatgrass juice and lifestyle recommendations on cancer patients' quality of life | 4 months
  Assessing impact of wheatgrass juice and lifestyle recommendations on cancer patients' quality of life(including fatigue)during chemotherapy

SECONDARY OUTCOMES:
Assessing compliance of patients to lifestyle recommendations during chemotherapy | 4 months
  Assessing compliance of patients to lifestyle recommendations (diet, physical activity and breathing exercises) during chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Eran Ben-Arye, MD, Principal Investigator — Clalait Health Services
Locations (1):
- Lin Medical Center, Haifa, Israel

REFERENCES:
- [Background] Bar-Sela G, Tsalic M, Fried G, Goldberg H. Wheat grass juice may improve hematological toxicity related to chemotherapy in breast cancer patients: a pilot study. Nutr Cancer. 2007;58(1):43-8. doi: 10.1080/01635580701308083. PMID 17571966